CLINICAL TRIAL: NCT00263458
Title: Integrating Buprenorphine Into the SFGH AIDS Program (Patient Evaluation Study)
Brief Title: Integrating Buprenorphine Into the SFGH AIDS Program
Acronym: BHIVES-SF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Department of Public Health (Other Government); The New York Academy of Medicine (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H97HA03799
Record Dates: First submitted 2005-12-06; First posted 2005-12-08 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: HIV; Buprenorphine; Opioid Dependence
Keywords: HIV; acquired immunodeficiency syndrome; buprenorphine; opioid dependence; opioid-related disorders; integrated care; primary care
MeSH Terms: conditions — Opioid-Related Disorders; Acquired Immunodeficiency Syndrome | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated (Experimental): Buprenorphine maintenance treatment delivered at an HIV primary care clinic
  Interventions: Other: Integrated office-based buprenorphine treatment for opioid dependence in an HIV primary care setting
- Non-integrated (Active Comparator): Buprenorphine maintenance treatment delivered at a public health substance use disorder clinic
  Interventions: Other: Integrated office-based buprenorphine treatment for opioid dependence in an HIV primary care setting

INTERVENTIONS:
Other: Integrated office-based buprenorphine treatment for opioid dependence in an HIV primary care setting — Eligible opioid-dependent HIV-infected patients are randomly assigned to receive buprenorphine opioid agonist treatment for 12 months either in an integrated HIV primary care setting (intervention group) versus a non-integrated substance use treatment clinic setting (comparison group).
  Other Names: Suboxone, Subutex

SUMMARY:
The purpose of this study is to assess the feasibility, cost, and effectiveness of a model of care designed to integrate buprenorphine treatment for opioid dependence into the HIV primary care clinics at the UCSF Positive Health Program.

DETAILED DESCRIPTION:
The UCSF Positive Health Program (formerly called the AIDS Program) at San Francisco General Hospital (SFGH) is one of the oldest and largest HIV/AIDS clinics in the United States. Located at the public hospital serving medically indigent residents of San Francisco, the Positive Health Program (PHP) provides over 2,000 patient visits per month to 2,300 patients in a comprehensive HIV primary care setting. The clinic population is disproportionately affected by heroin and other opiate abuse problems. Opiate replacement therapy (ORT) has a stabilizing effect in HIV-infected injecting drug users (IDU) and is associated with greater acceptance of antiretroviral (ARV) therapy, higher ARV adherence, and greater engagement in appropriate HIV-related health care. However, there are insufficient resources to meet the critical substance abuse treatment needs among our opioid-dependent patients.

In partnership with the Community Behavioral Health Services (CBHS) section of the San Francisco Department of Public Health (SFDPH), the UCSF Positive Health Program (PHP) at San Francisco General Hospital (SFGH) has developed a model of care, which provides opioid-dependent patients with integrated, office-based buprenorphine ORT in the HIV primary care setting. The program also offers primary care providers with education and training on addiction, opiate addiction treatment, and the appropriate use of buprenorphine. An evaluation of the program is planned to examine: (1) its effects on the health and substance use of patients; (2) program costs; and (3) what broader impact the program has on providers, institutions, and local systems. In the patient evaluation study, eligible, opioid-dependent patients that receive primary HIV care at the PHP will be randomly assigned to receive buprenorphine ORT for twelve months either in the integrated HIV primary care setting (intervention group) versus a non-integrated substance abuse treatment clinic setting (comparison group). Data will be abstracted from medical chart reviews and will be collected from patients using standardized instruments and satisfaction surveys.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Fluent in English
* Receive HIV primary care at the UCSF Positive Health Program
* Meet DSM-IVR criteria for opioid dependence
* Meet clinical criteria for buprenorphine treatment (see Exclusion Criteria)
* Plan to stay in the San Francisco Bay Area for the next 12 months

Exclusion Criteria:

* Severe hepatic dysfunction, i.e., AST and/or ALT > 5X upper limit of normal
* DSM-IV criteria for benzodiazepine abuse or dependence within the past 6 months
* DSM-IV criteria for alcohol dependence within the past 6 months
* Actively suicidal
* Psychiatric impairment that impedes ability to consent (dementia, delusional, actively psychotic)
* Methadone or opiate analgesic doses exceed level allowing for safe transition to buprenorphine
* Pregnant women and women actively trying to become pregnant

Potential subjects also will be excluded for:

* Any medical condition(s), which, in the opinion of the investigator, would interfere with the patient's ability to participate in or adhere to the requirements of this study
* Unable or who decline to provide informed consent for the evaluation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Substance use outcomes at 0, 1, 3, 6, 9 and 12 months. | 0, 1, 3, 6, 9 and 12 months.
HIV care outcomes at 0, 1, 3, 6, 9 and 12 months. | 0, 1, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
HIV-related health | baseline, 1, 3, 6, 9 and 12 months
Quality of life | 0, 1, 3, 6, 9 and 12 months
Social functioning | 0, 1, 3, 6, 9 and 12 months
Quality of HIV care. | 0, 3, 6, 9 and 12 months
Patient satisfaction at 3 months. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Paula J Lum, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Positive Health Program, San Francisco, California, United States

REFERENCES:
- [Result] Korthuis PT, Fiellin DA, Fu R, Lum PJ, Altice FL, Sohler N, Tozzi MJ, Asch SM, Botsko M, Fishl M, Flanigan TP, Boverman J, McCarty D; BHIVES Collaborative. Improving adherence to HIV quality of care indicators in persons with opioid dependence: the role of buprenorphine. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1(Suppl 1):S83-90. doi: 10.1097/QAI.0b013e31820bc9a5. PMID 21317600
- [Result] Sullivan LE, Botsko M, Cunningham CO, O'Connor PG, Hersh D, Mitty J, Lum PJ, Schottenfeld RS, Fiellin DA; BHIVES Collaborative. The impact of cocaine use on outcomes in HIV-infected patients receiving buprenorphine/naloxone. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1(Suppl 1):S54-61. doi: 10.1097/QAI.0b013e3182097576. PMID 21317595
- [Result] Fiellin DA, Weiss L, Botsko M, Egan JE, Altice FL, Bazerman LB, Chaudhry A, Cunningham CO, Gourevitch MN, Lum PJ, Sullivan LE, Schottenfeld RS, O'Connor PG; BHIVES Collaborative. Drug treatment outcomes among HIV-infected opioid-dependent patients receiving buprenorphine/naloxone. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1(0 1):S33-8. doi: 10.1097/QAI.0b013e3182097537. PMID 21317592
- [Result] Altice FL, Bruce RD, Lucas GM, Lum PJ, Korthuis PT, Flanigan TP, Cunningham CO, Sullivan LE, Vergara-Rodriguez P, Fiellin DA, Cajina A, Botsko M, Nandi V, Gourevitch MN, Finkelstein R; BHIVES Collaborative. HIV treatment outcomes among HIV-infected, opioid-dependent patients receiving buprenorphine/naloxone treatment within HIV clinical care settings: results from a multisite study. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1(Suppl 1):S22-32. doi: 10.1097/QAI.0b013e318209751e. PMID 21317590
- [Result] Vergara-Rodriguez P, Tozzi MJ, Botsko M, Nandi V, Altice F, Egan JE, O'Connor PG, Sullivan LE, Fiellin DA; BHIVES Collaborative. Hepatic safety and lack of antiretroviral interactions with buprenorphine/naloxone in HIV-infected opioid-dependent patients. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1:S62-7. doi: 10.1097/QAI.0b013e31820a820f. PMID 21317596
- [Result] Weiss L, Netherland J, Egan JE, Flanigan TP, Fiellin DA, Finkelstein R, Altice FL; BHIVES Collaborative. Integration of buprenorphine/naloxone treatment into HIV clinical care: lessons from the BHIVES collaborative. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1:S68-75. doi: 10.1097/QAI.0b013e31820a8226. PMID 21317597
- [Result] Finkelstein R, Netherland J, Sylla L, Gourevitch MN, Cajina A, Cheever L; BHIVES Collaborative. Policy implications of integrating buprenorphine/naloxone treatment and HIV care. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1:S98-S104. doi: 10.1097/QAI.0b013e31820a9a97. PMID 21317602
- [Result] Chaudhry AA, Botsko M, Weiss L, Egan JE, Mitty J, Estrada B, Lucas GM, Woodson T, Flanigan TP, Fiellin DA; BHIVES Collaborative. Participant characteristics and HIV risk behaviors among individuals entering integrated buprenorphine/naloxone and HIV care. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1:S14-21. doi: 10.1097/QAI.0b013e318209d3b9. PMID 21317589
- [Result] Weiss L, Egan JE, Botsko M, Netherland J, Fiellin DA, Finkelstein R. The BHIVES collaborative: organization and evaluation of a multisite demonstration of integrated buprenorphine/naloxone and HIV treatment. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1:S7-13. doi: 10.1097/QAI.0b013e3182097426. PMID 21317598
- [Result] Cheever LW, Kresina TF, Cajina A, Lubran R. A model federal collaborative to increase patient access to buprenorphine treatment in HIV primary care. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1:S3-6. doi: 10.1097/QAI.0b013e318209740f. PMID 21317591
- [Result] Friedland G, Vlahov D. Integration of buprenorphine for substance-abuse treatment by HIV care providers. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1:S1-2. doi: 10.1097/QAI.0b013e31820bc9ba. No abstract available. PMID 21317588
- See also: The UCSF Positive Health Program at the University of California San Francisco — http://php.ucsf.edu/
- See also: Integrated Buprenorphine & HIV Care Evaluation and Support Center — http://www.bhives.org/
- See also: Community Behavioral Health Services, San Francisco Department of Public Health — http://www.sfdph.org/dph/comupg/oservices/mentalHlth/CBHS/default.asp
- See also: JAIDS. March 1, 2011 - Volume 56 - Supplement 1, Integration of Buprenorphine/Naloxone Treatment into HIV Clinical Care — http://journals.lww.com/jaids/toc/2011/03011